CLINICAL TRIAL: NCT04818528
Title: Effects of Constraint Induced Movement Therapy on Hand and Arm Functions in Patients of Parkinson's Disease
Brief Title: Effects of CIMT in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: Riphah International University (Other)
Responsible Party: Principal Investigator, Mariam Ghazanfar, Senior Lecturer, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/20/0214
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Constraint induced movement therapy; Upper limb; Physical therapy; Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: It was a parallel group, randomized controlled trial of 40 Parkinson's disease patients enrolled between December 2020 to Feb 2021.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint Induced Movement Therapy and Routine Physical Therapy (Experimental): Patients received constrained induced movement therapy and routine physical therapy for up to 6 hrs/day, 5 days/week for 4 weeks.
  Interventions: Other: Constraint Induced Movement Therapy and Routine Physical Therapy
- Routine Physical Therapy (Active Comparator): Patients received routine physical therapy for 5 days/week for 4 weeks.
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Constraint Induced Movement Therapy and Routine Physical Therapy — Intensive, graded practice of the paretic upper limb to enhance task-specific use of the affected limb. Constraint or forced use therapy, with the non-paretic upper limb contained in a mitt to promote the use of the impaired limb during 90% of the total hours awake. Adherence enhancing behavioral methods designed to transfer the gains obtained in the clinical setting or the laboratory to patients' real-world environment (ie, a transfer package).
  As part of routine physical therapy patients received intervention that worked on aerobic capacity, muscle strengthening exercise, walking ability, postural and balance disorders and improving hand arm function. Three stages were used in each session: (i) warm-up phase: passive mobilization of major joints and lower limb muscle strengthening; (ii) active phase (both standing and sitting): motor control exercises for upper and lower limbs, and (iii) cool down phase (in seating position): respiratory exercises and mobilization.
  Arms: Constraint Induced Movement Therapy and Routine Physical Therapy
Other: Routine Physical Therapy — As part of routine physical therapy patients received intervention that worked on aerobic capacity, muscle strengthening exercise, walking ability, postural and balance disorders and improving hand arm function. Three stages were used in each session: (i) warm-up phase: passive mobilization of major joints and lower limb muscle strengthening; (ii) active phase (both standing and sitting): motor control exercises for upper and lower limbs, and (iii) cool down phase (in seating position): respiratory exercises and mobilization.
  Arms: Routine Physical Therapy

SUMMARY:
The purpose of the study was to determine the effects of constraint induced movement therapy on hand and arm functions in Parkinson's disease patients. It was a randomized controlled trial, conducted in physical therapy department of University of Lahore Teaching Hospital, Mayo Hospital and Lahore General Hospital. 40, male and female Parkinson's disease patients aged between 50-80 years were randomly allocated into two equal groups. In experimental group patients were treated with constraint induced movement therapy and routine physical therapy and in control group patients were treated with routine physical therapy. Patients were treated for a total of 4 weeks, 6 hours in a day. Patients were assessed using Frenchay Arm Test (FAT). SPSS 25 was used to analyze the data.

DETAILED DESCRIPTION:
One of the central nervous system's most frequent diseases is Parkinson's disease (PD). In individuals with PD upper limb impairments could be present such as resting tremor or micrographia, often the first symptom of the disorder. These upper limb conditions can lead to difficulties in work, leisure, and everyday activities such as eating and dressing as the disease advances. This research was aimed to provide insightful information for both clinicians, researchers and for community in general. This study was helpful in the field of neurorehabilitation to bridge the gaps of previous researches. Clinician or neurorehabilitation expert can apply the more useful technique on patients and get the better results in less time. Researchers can find the high-quality clinical evidence regarding constraint induced movement therapy on Parkinson's patients. According to evidence-based practice patient preference is considered in providing treatments to patients. So, patient can find out which treatment is better.

40 patients who fulfill the inclusion criteria were enrolled in this study. Written informed consent was taken from every subject participating in this study. Allocation of subjects in two groups was done by random number table. Group A was treated with Constrained Induced movement therapy along with routine physical therapy and group B was treated only with routine physical therapy. In routine physical therapy group patients received intervention according to systematic review and clinical guidelines that worked on aerobic capacity, muscle strengthening exercise, walking ability, postural and balance disorders and improving hand arm function.39 Three stages were used in each session: (i) warm-up phase: passive mobilization of major joints and lower limb muscle strengthening; (ii) active phase (both standing and sitting): motor control exercises for upper and lower limbs, and (iii) cool-down phase (in seating position): respiratory exercises and mobilization.

40 The routine or baseline therapy was remained same throughout the study. Constraint induced movement therapy was given to group A for four weeks. Training was done for 6 hrs/day, 5 days/week for 4 weeks. All the information wascollected by using standardized questionnaire of Frenchay arm test. Confounding variables were controlled by randomization and restriction methods. All treatment was given by single therapist to control the biasness.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's disease referred from neurology department.
* Parkinson's disease patients with age range 50- 80 years.
* Both male and female patients.

Exclusion Criteria:

* Atypical Parkinsonism Alzheimer's disease
* Any patient taking antidepressants other than Parkinson's
* Patients of severe cognitive impairments.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Frenchay Arm Test | Change from Baseline at 4 weeks
  The Frenchay Arm Test (FAT) is a measure of upper extremity proximal motor control and dexterity during ADL performance in patients with impairments of upper extremity resulting from neurological conditions. FAT is an upper extremity specific measure of activity limitation. The Frenchay Arm Test is an ordinal 2-point scale (0-1). 0 for fail and 1 for pass. A total of 5 points can be obtained (range 0-5) with better score demonstrating better performance. FAT took about 3 minutes to administer.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Ghazanfar, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No